CLINICAL TRIAL: NCT02835378
Title: Observational Study of Bilateral Upper Limb Amputees in France
Brief Title: Bilateral Upper Limb Amputation Observatory
Acronym: ARMOBS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0465
Record Dates: First submitted 2016-07-13; First posted 2016-07-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Bilateral Upper Limb Amputation; Transverse Short Amputation of the Hand; Arm Amputation
Keywords: bilateral upper limb amputation; prosthetic fitting; epidemiology; clinical practices; totally non-functional hand

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bilateral upper limb amputation: Bilateral upper limb amputees, with amputation from the short transverse hand (hand completely non-functional) to complete arm, whatever their age
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
In France, there is currently no data to directly estimate the number of bilateral upper limb amputations, their characteristics and therapeutic care.

By extrapolation from the Regional Institute of Physical Medicine and Rehabilitation (PMR) Nancy in 2005, the number of new cases of amputated patients with prosthetic fitting of the upper limb was estimated at 355. Epidemiological data from the 2009-2010 Annual Report of the LIMBLESS STATISTICS database (collection of quantitative clinical data and demographic of amputees patients referred by orthopaedic centres in the United Kingdom , whose population's characteristics are similar to France) identified 395 incident cases of upper limb amputation with, 6 bilateral amputations observed. The causes are varied: traumatic, infectious or related to diabetes. The population was relatively young, aged between 15 and 54 year old.

On this basis, the estimated number of new cases of bilateral upper limb amputations throughout France should therefore be about 40 incident cases over a 5-year period.

This observational study is aimed at collecting comprehensive and high quality data to describe the French population of bilateral upper limb amputees.

ELIGIBILITY:
Inclusion Criteria:

All French patients :

* presenting bilateral upper limb amputation, from short transverse amputation of the hand (hand not fully functional) to arm amputation;
* affiliated with a social security scheme or assimilated;
* who have given their non-opposition to participate in the study.

Exclusion Criteria:

* Patients with finger amputation only;
* Patients already having prosthesis of one upper limb (first amputation) and willing to receive prosthesis fitting after a contralateral amputation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All incident case of bilateral upper limb amputation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-12; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Etiology of amputation | At the time of the bilateral amputation (Day 0)
  Etiological characteristics of bilateral upper limb amputees
Amputation level on each side | At the time of the bilateral amputation (Day 0)
  Epidemiological characteristics of bilateral upper limb amputees

SECONDARY OUTCOMES:
Number and indication of surgical interventions | At the time the stumps are healed (an average of 1 month)
Number and type of surgical and medical complications | At the time the stumps are healed (an average of 1 month)
Length of stay in the hospital | At the time the stumps are healed (an average of 1 month)
Duration before entry into rehabilitation centre | At the time the stumps are healed (an average of 1 month)
Duration from surgical amputation to healing of the stumps | At the time the stumps are healed (an average of 1 month)
Duration from surgical amputation to prosthesis fitting | At the time the stumps are healed (an average of 1 month)
Type of planned prosthesis | At the time the stumps are healed (an average of 1 month)

CONTACTS AND LOCATIONS:
Overall Officials: Lionel BADET, Pr, Principal Investigator — Hospices Civils de Lyon, Hôpital Edouard Herriot
Locations (1):
- Hospices Civils de Lyon, Hôpital Edouard Herriot, Lyon, France